CLINICAL TRIAL: NCT03025802
Title: Fast Assay for Pathogen Identification and Characterization - Prospective Study
Acronym: FAPIC
Status: Completed | Type: Observational
Sponsor: Hasselt University (Other)
Collaborators: AIT Austrian Institute of Technology GmbH (Other); University of Zagreb (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, prof. dr. Inge Gyssens, Prof. dr., Hasselt University
Other Study IDs: 16.120/infect16.04
Record Dates: First submitted 2017-01-13; First posted 2017-01-20 (Estimated); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Sepsis
Keywords: Molecular diagnosis; Pathogen identification; Sepsis; Bacteremia; Rapid diagnostics
MeSH Terms: conditions — Sepsis; Bacteremia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The FAPIC project will develop a diagnostic system that will identify pathogens and charachterize virulence and resistance. A prospective study will be performed in which blood samples will be collected of patients with suspected sepsis in order to evaluate the diagnostic system. In routine care, blood is drawn of these patients for culture in order to identify the causative pathogen. This process takes 3-5 days. During the study, one extra blood sample will be collected with the same venipuncture, with each blood culture. Afterwards, routine diagnosis by blood culture is followed. Blood samples will be send to the research laboratories for determination of sensitivity and specificity. The system will not be used in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Suspicion of bacteremia

Exclusion Criteria:

* Children (<18 years)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective cohort will be set up to determine and evaluate the performance of the diagnostic system. The cohort will consist of 250 patients (~500 blood culture sets) with suspicion of bacteremia, for whom routine blood cultures are ordered.
Sampling Method: Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Detection of pathogens and its virulence factors and susceptibility genes | 1 year
  Sensitivity, specificity, and accuracy of the molecular system compared to blood culture.

SECONDARY OUTCOMES:
Population outcome during routine procedures | 1 year
  Insights on routine hospital procedures using blood culture and outcomes on the study population such as TAT, antimicrobial use, time to antimicrobial change, in-hospital stay, and mortality by collection of patient data in the medical records.

CONTACTS AND LOCATIONS:
Overall Officials: Inge C Gyssens, MD, PhD, Principal Investigator — Hasselt University
Locations (2):
- Jessa Hospital, Hasselt, Limburg, Belgium
- University of Zagreb Medical School, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Martin GS. Sepsis, severe sepsis and septic shock: changes in incidence, pathogens and outcomes. Expert Rev Anti Infect Ther. 2012 Jun;10(6):701-6. doi: 10.1586/eri.12.50. PMID 22734959
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb S, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including The Pediatric Subgroup. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock, 2012. Intensive Care Med. 2013 Feb;39(2):165-228. doi: 10.1007/s00134-012-2769-8. Epub 2013 Jan 30. PMID 23361625
- [Background] Yoshikawa TT. Antimicrobial resistance and aging: beginning of the end of the antibiotic era? J Am Geriatr Soc. 2002 Jul;50(7 Suppl):S226-9. doi: 10.1046/j.1532-5415.50.7s.2.x. PMID 12121517
- [Background] Corona A, Colombo R. Towards the end of the antibiotic era: let's save the ancient soldier Colistin! Intensive Care Med. 2013 Sep;39(9):1660-1. doi: 10.1007/s00134-013-2955-3. Epub 2013 May 22. No abstract available. PMID 23695267
- [Background] Hede K. Antibiotic resistance: An infectious arms race. Nature. 2014 May 1;509(7498):S2-3. doi: 10.1038/509S2a. No abstract available. PMID 24784426
- [Background] Bush K. Alarming beta-lactamase-mediated resistance in multidrug-resistant Enterobacteriaceae. Curr Opin Microbiol. 2010 Oct;13(5):558-64. doi: 10.1016/j.mib.2010.09.006. Epub 2010 Oct 1. PMID 20920882
- [Background] Zankari E, Hasman H, Cosentino S, Vestergaard M, Rasmussen S, Lund O, Aarestrup FM, Larsen MV. Identification of acquired antimicrobial resistance genes. J Antimicrob Chemother. 2012 Nov;67(11):2640-4. doi: 10.1093/jac/dks261. Epub 2012 Jul 10. PMID 22782487
- See also: FAPIC project website — http://www.fapic.eu